CLINICAL TRIAL: NCT03277469
Title: Optimizing Brachytherapy Application and Delivery With MRI Guidance for Gynecologic Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Martin King, MD, PhD, Associate Professor of Radiation Oncology, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-128
Record Dates: First submitted 2017-09-07; First posted 2017-09-11 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Gynecologic Cancer
Keywords: Gynecologic Cancer
MeSH Terms: interventions — Brachytherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- MRI Guided BRACHYTHERAPY with Tracker (Experimental): * Standard pelvic MRI sequences will be obtained
  * MRI Tracker is used during catheter positioning with serial MR imaging during implant
  * All patients will undergo 3D-based image acquisition for brachytherapy treatment planning per standard clinical practice
  * The brachytherapy modality to be used is high-dose-rate brachytherapy using an iridum-192 stepping source
  Interventions: Device: MRI; Radiation: Brachytherapy; Device: MRI Tracker
- MRI Guided BRACHYTHERAPY without Tracker (Experimental): * Standard pelvic MRI sequences will be obtained
  * Standard process is used with serial MR imaging to evaluate catheter position during implant
  * All patients will undergo 3D-based image acquisition for brachytherapy treatment planning per standard clinical practice
  * The brachytherapy modality to be used is high-dose-rate brachytherapy using an iridum-192 stepping source
  Interventions: Device: MRI; Radiation: Brachytherapy

INTERVENTIONS:
Device: MRI — Medical imaging technique used in radiology to form pictures of the anatomy and the physiological processes of the body
Radiation: Brachytherapy — Radiation therapy that is delivered by inserting radioactive sources directly into a tumor
Device: MRI Tracker — The MR tracking device consists of a series of radiofrequency (RF) microcoils that are embedded into brachytherapy catheter stylet. The RF microcoils allows for accurate spatial localization of an individual brachytherapy catheter.
  Arms: MRI Guided BRACHYTHERAPY with Tracker

SUMMARY:
The aim of this study is to develop new tools using magnetic resonance imaging (MRI) that will improve the brachytherapy procedure and treatment for participants with gynecologic cancer.

DETAILED DESCRIPTION:
This research study is designed to develop new technology using MR imaging to improve the brachytherapy procedure for participants with gynecologic cancer. The brachytherapy procedure will take place in an MRI procedure room within the Advanced Multimodality Image-Guided Operating (AMIGO) suite at Brigham and Women's Hospital. The purpose of the study will be to evaluate whether the use of an MR-tracking device will improve the placement of the brachytherapy catheters. This information will also be used to develop new software for real-time brachytherapy planning by our physics team. The investigators believe that the development of an MR-tracking device will allow them to better place the brachytherapy catheters for radiation treatment and ultimately improve outcomes for patients, including better local tumor control and a lower risk of side effects. The investigators will also evaluate new MRI protocols to better define the tumor at the time of brachytherapy. The brachytherapy treatment planning and delivery will follow standard of care.

In the past, brachytherapy treatment planning and delivery for gynecologic cancer was based on plain-film X-rays, which did not account for the shape of the tumor, the unique anatomy of an individual patient or the response to pelvic radiation therapy. In the last decade, advances in technology have made it possible to perform the brachytherapy procedure and to plan the delivered radiation dose based on CT or MR imaging. The use of CT or MR imaging for brachytherapy planning is increasingly common in the United States, and has been shown to result in improved tumor controls rates and a lower risk of radiation complications. The use of MRI-guidance during the brachytherapy procedure is unique and this study will contribute the advancement of this important technology. About half of the participants in this study will be selected to have the MRI-guided brachytherapy procedure with the use of an MRI-tracking device. This device will provide real-time positioning information of the individual brachytherapy catheters while they are being placed and adjusted within the tumor. The MR-tracker will also be used to develop new software that will allow our physics team to generate a near-instantaneous brachytherapy plan as individual catheters are placed during the procedure. The investigators hope that these advances in technology will have a meaningful impact on further increasing tumor control and limiting the complication risk for our participants.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and the willingness to sign a written informed consent document. Subject is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.
* Participants must have a biopsy-proven diagnosis of primary or recurrent gynecologic cancer for which intracavitary or interstitial brachytherapy is planned as standard treatment. Eligible disease sites include primary or recurrent cancer of endometrial, ovarian, cervical, vaginal, or vulvar origin.
* Age of 18 years or older are eligible.
* ECOG performance status of 2 or less.
* Patients who have received prior radiation or chemotherapy may be enrolled on this study.
* Participant is deemed to be an appropriate candidate for MRI-guided brachytherapy by the radiation oncologist and the patient elects to be treated with MRI-guided brachytherapy.
* Participant provides informed consent for prospective collection of relevant medical records for analysis of clinical outcome and treatment-planning techniques.

Exclusion Criteria:

* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, uncontrolled hypertension, interstitial lung disease, active peptic ulcer disease or gastritis, active bleeding diatheses, serious chronic gastrointestinal conditions associated with diarrhea or psychiatric illness/social situations that would limit compliance with study requirements.
* Contraindication to MRI identified by the MR procedure screening form, such as a pacemaker, aneurysm clip, inner ear implant, neurostimulator, or other non-MR compatible implant or device.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2017-11-13 (Actual); Primary Completion 2025-09-15 (Estimated); Study Completion 2027-09-15 (Estimated)

PRIMARY OUTCOMES:
Brachytherapy treatment parameters, including V150 | 3 weeks
  Comparison of brachytherapy treatment parameters for patients treated with or without use of an MR-tracker. V150 is the tumor volume that receives at least 150% of the prescribed radiation dose and is a measure of radiation dose heterogeneity

SECONDARY OUTCOMES:
Local-Failure-Free Survival | Baseline to 2 years, 5 years
  Time from diagnosis or recurrence to time of local failure
Progression Free Survival | Baseline to 2 years, 5 years
  Time from diagnosis or recurrence to time of documented progression or death
Overall Survival | Baseline to 2 years, 5 years
  Time from diagnosis or recurrence to time of death

CONTACTS AND LOCATIONS:
Overall Officials: Martin King, MD, PhD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No